CLINICAL TRIAL: NCT00496119
Title: Phase II Evaluation of Proton Beam Therapy for Skull Base Chordoma
Brief Title: Proton Beam Therapy for Chordoma Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0038; NCI-2012-01509 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chordoma
Keywords: Proton Beam Therapy; Skull Base Chordoma; Chordoma of the Skull Base; Chordoma
MeSH Terms: conditions — Chordoma | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- 70 Gray (Gy) Proton Beam Therapy (Experimental): Participants treated to 70 cobalt Gray equivalent (CGE) only (the standard treatment).
  Interventions: Radiation: Proton Beam Therapy
- Photon Beam Therapy (Experimental): Proton beam therapy combined with photon radiation therapy where combination improves final dose distribution.
  Interventions: Radiation: Proton Beam Therapy; Radiation: Photon Beam Therapy

INTERVENTIONS:
Radiation: Proton Beam Therapy — 70 Gy once daily at 2 CGE per fraction, no sooner than 2 weeks after last surgery to remove tumor, for between 35-39 treatments.
Radiation: Photon Beam Therapy — Photon beam therapy once daily, no sooner than 2 weeks after last surgery to remove tumor, for 35-39 treatments.
  Arms: Photon Beam Therapy

SUMMARY:
The goal of this clinical research study is to learn if proton beam therapy, with or without photon beam radiation therapy, is effective in the treatment of skull base chordoma. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Proton therapy is a kind of external beam radiation therapy where protons are directed to a tumor site. Researchers are trying to determine what level of proton therapy gives the most benefit without causing toxic side effects. Researchers will also be testing the treatment's effect.

If your doctor feels it is necessary, the proton beam therapy may be combined with standard photon therapy.

If you are eligible to take part in this study, you will receive proton beam therapy at The University of Texas (UT) MD Anderson Cancer Center (MDACC), and possibly photon beam, no sooner than 2 weeks after the last surgery to remove the tumor. You will receive proton beam therapy once a day for about 35 treatments (7 weeks). Treatment will be given for 5 days in a row each week (except for Saturdays, Sundays and holidays) at the MDACC Proton Center in Houston. The whole process should take up to 1 hour each day.

This is an investigational study. The proton beam machine used to deliver treatment is approved by the FDA for patient use. The doses being studied are experimental. About 15 participants will take part in this study. All will be enrolled at MDACC.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed chordoma of the skull base
2. Contrast enhanced postoperative MRI (CT in case MRI is contraindicated) of the skull base obtained within 90 days of study registration
3. MDACC surgeons have determined that optimal debulking of disease has been performed.
4. Karnofsky Performance status greater than or equal to 60
5. Signed informed consent

Exclusion Criteria:

1. Previous irradiation of the skull base
2. Documented evidence of disseminated metastatic disease
3. Any concurrent malignancy (other than non-melanoma skin cancers) in the last 3 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-09-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to Local Recurrence | 1 year after radiation treatments
  Recurrence classified as "central," "in-field", "marginal," "peripheral," or "distant" depending upon its relationship to the dose distribution on the original treatment plan.
  MRI (or CT in case MRI is contraindicated) of the skull base used to document the status of disease in the following categories: 1) stable disease, 2) progressive disease, 3) partial response/complete response. A post-operative MRI (or CT) obtained within 90 days of study registration serves as baseline with annual follow up till disease progression or death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: David Grosshans, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org